CLINICAL TRIAL: NCT02597049
Title: A Randomized, Parallel-Arm, Double-Blind Study of Efficacy and Safety of Dulaglutide When Added to SGLT2 Inhibitors in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of Dulaglutide (LY2189265) in Participants With Type 2 Diabetes Mellitus
Acronym: AWARD-10
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15361; H9X-MC-GBGE (Other: Eli Lilly and Company); 2015-002095-24 (EudraCT Number)
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Sodium-Glucose Transporter 2 Inhibitors; Canagliflozin; dapagliflozin; empagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1.5 mg Dulaglutide (Experimental): 1.5 milligrams (mg) given subcutaneously (SC) once a week for 24 weeks.
  Interventions: Drug: Dulaglutide; Drug: SGLT2 inhibitor; Drug: Metformin
- 0.75 mg Dulaglutide (Experimental): 0.75 mg dulaglutide given SC once a week for 24 weeks.
  Interventions: Drug: Dulaglutide; Drug: SGLT2 inhibitor; Drug: Metformin
- Placebo (Placebo Comparator): Placebo given SC once a week for 24 weeks.
  Interventions: Drug: Placebo; Drug: SGLT2 inhibitor; Drug: Metformin

INTERVENTIONS:
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
  Arms: 0.75 mg Dulaglutide; 1.5 mg Dulaglutide
Drug: Placebo — Administered SC
  Arms: Placebo
Drug: SGLT2 inhibitor — Administered orally as standard of care for type 2 diabetes
  Other Names: Canagliflozin; Dapagliflozin; Empagliflozin
Drug: Metformin — Administered orally as standard of care for type 2 diabetes

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of the study drug known as dulaglutide when added to sodium-glucose co-transporter 2 (SGLT2) inhibitors in participants with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus (based on the World Health Organization's [WHO] diagnostic criteria)
* Have been treated with an SGLT2 inhibitor, with or without metformin, for at least 3 months prior to study entry (minimum required doses for that period for allowed SGLT2 inhibitors: empagliflozin 10 mg, dapagliflozin 5 or 10 mg [per country-specific label], canagliflozin 100 mg); minimum required dose for metformin, if used, is ≥1500 mg/day and must be reached (or highest tolerated dose which is acceptable with documented gastrointestinal [GI] intolerability)
* Daily doses of all allowed oral antihyperglycemia agent (OAMs) must have been stable for at least 12 weeks (±3 days) prior to randomization (study enrollment); daily doses of SGLT2 inhibitor and metformin, if used, will be considered stable during this period if:

  * all prescribed daily doses were in the range between the minimum required dose and maximum-approved dose per country-specific label; and
  * >90% of prescribed daily doses were equal to the dose at randomization
* Have HbA1c ≥7.0% and ≤9.5% at study entry and approximately 1 week prior to randomization
* Have body mass index (BMI) ≤45 kilograms per meter squared (kg/m^2) and agree to not initiate a diet and/or exercise program during the study with the intent of reducing body weight other than the lifestyle and dietary measures for diabetes treatment

Exclusion Criteria:

* Have type 1 diabetes mellitus
* Have been treated with any other OAMs (other than SGLT2 inhibitors and metformin), glucagon-like peptide-1 receptor agonist (GLP-1 RA), pramlintide or insulin 3 months prior to study entry, or between study entry and randomization; or initiate metformin between study entry and randomization; short-term use of insulin for acute care (≤14 days) during the 3-month period prior to entry is not exclusionary
* Have any condition that is a contraindication for use of the GLP-1 RA class or the SGLT2 inhibitor class (per country-specific labels) at study entry or develop such condition between study entry and randomization
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease other than nonalcoholic fatty liver disease (NAFLD), or alanine transaminase (ALT) level >2.5 times the upper limit of the reference range, as determined by the central laboratory at study entry; participants with NAFLD are eligible for participation in this trial
* Had chronic or acute pancreatitis any time prior to study entry
* Estimated glomerular filtration rate (eGFR) <45 milliliters(mL)/minute/1.73m^2, calculated by the Chronic Kidney Disease-Epidemiology (CKD-EPI) equation, as determined by the central laboratory at study entry and confirmed at lead in
* Have any self or family history of type 2A or type 2B multiple endocrine neoplasia (MEN 2A or 2B) in the absence of known C-cell hyperplasia (this exclusion includes participants with a family history of MEN 2A or 2B, whose family history for the syndrome is rearranged during transfect [RET]-negative; the only exception for this exclusion will be for participants whose family members with MEN 2A or 2B have a known RET mutation and the potential participant for the study is negative for the RET mutation)
* Have any self or family history of medullary C-cell hyperplasia, focal hyperplasia, carcinoma (including sporadic, familial, or part of MEN 2A or 2B syndrome)
* Have a serum calcitonin ≥20 picograms/mL as determined by the central laboratory at study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- United States (13):
  - Medical Group of Encino, Encino, California
  - National Research Institute, Huntington Park, California
  - National Research Institute, Los Angeles, California
  - New Horizon Research Center, Miami, Florida
  - Metabolic Research Institute Inc., West Palm Beach, Florida
  - Cotton O'Neil Diabetes and Endocrinology Center, Topeka, Kansas
  - JCMG Clinical Research, Jefferson City, Missouri
  - Grand Street Medical PC, Brooklyn, New York
  - Diabetes & Endocrinology Consultants PC, Morehead City, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - Galenos Research, Dallas, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
- Austria (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Stefan Ob Stainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Steyr
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Czechia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Brandys Nad Labem-Stara Bolesl
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holešov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krnov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pardubice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oldenburg
- Hungary (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagykanizsa
- Israel (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zapopan
- Puerto Rico (3):
  - Centro de Endocrinologia y Nutricion, Caguas
  - Manati Medical Center, Manatí
  - Centro de Endocrinologia del Este, Yabucoa
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Ferdinand KC, Dunn J, Nicolay C, Sam F, Blue EK, Wang H. Weight-dependent and weight-independent effects of dulaglutide on blood pressure in patients with type 2 diabetes. Cardiovasc Diabetol. 2023 Mar 9;22(1):49. doi: 10.1186/s12933-023-01775-x. PMID 36894938
- [Derived] Ludvik B, Frias JP, Tinahones FJ, Wainstein J, Jiang H, Robertson KE, Garcia-Perez LE, Woodward DB, Milicevic Z. Dulaglutide as add-on therapy to SGLT2 inhibitors in patients with inadequately controlled type 2 diabetes (AWARD-10): a 24-week, randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2018 May;6(5):370-381. doi: 10.1016/S2213-8587(18)30023-8. Epub 2018 Feb 23. PMID 29483060
- See also: Click here for more information about this study: A Study of Dulaglutide (LY2189265) in Participants With Type 2 Diabetes Mellitus — http://www.lillytrialguide.com/EN-US/studies/diabetes/gbge

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.5 mg Dulaglutide: Dulaglutide 1.5 milligrams (mg) given SC QW for 24 weeks.
- 0.75 mg Dulaglutide: Dulaglutide 0.75 mg given subcutaneously (SC) once a week (QW) for 24 weeks.
- Placebo: Placebo given SC QW for 24 weeks.
Period: Overall Study
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Placebo
Started | 142 | 142 | 140
Received at Least One Dose of Study Drug | 142 | 141 | 140
Completed | 135 | 137 | 137
Not Completed | 7 | 5 | 3
Not completed — Lost to Follow-up | 0 | 3 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Noncompliant with Study Visits | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Placebo | Total
Number analyzed (Participants) | 142 | 141 | 140 | 423
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.17 (9.26) | 58.55 (9.14) | 57.10 (9.59) | 57.27 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 72 | 74 | 211
  Male | 77 | 69 | 66 | 212
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 44 | 44 | 139
  Not Hispanic or Latino | 90 | 97 | 94 | 281
  Unknown or Not Reported | 1 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 4 | 7
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 6 | 12
  White | 127 | 127 | 124 | 378
  More than one race | 11 | 8 | 6 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 9 | 11 | 9 | 29
  Hungary | 19 | 19 | 19 | 57
  United States | 30 | 30 | 28 | 88
  Czechia | 25 | 23 | 25 | 73
  Mexico | 27 | 28 | 28 | 83
  Israel | 6 | 6 | 6 | 18
  Germany | 12 | 11 | 10 | 33
  Spain | 14 | 13 | 15 | 42
Baseline Mean Hemoglobin A1c (HbA1c) Treatment-Regimen Estimand [Mean (Standard Deviation); unit: percentage of HbA1c] — Population: All randomized participants who received at least one dose of study drug and had a baseline measure of HbA1c.
  percentage of HbA1c
    number analyzed (Participants) | 140 | 139 | 137 | 416
    (all) | 8.04 (0.66) | 8.04 (0.61) | 8.05 (0.66) | 8.04 (0.64)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at 24 Weeks (Treatment-regimen Estimand)
Description: Least Squares mean (LS) of the HbA1c change from baseline to primary endpoint at week 24 was adjusted by treatment, country, SGLT2 inhibitor dose, metformin use, treatment-by-visit interactions as fixed effects, and baseline HbA1c as a covariate and participant as a random effect, via a MMRM analysis. The treatment-regimen estimand used all data including post-rescue data and compared the benefit of treatment regimens as they were actually taken.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study medication and had evaluable data.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- 1.5 mg Dulaglutide: Dulaglutide 1.5 mg given SC QW for 24 weeks.
- 0.75 mg Dulaglutide: Dulaglutide 0.75 milligrams (mg) given subcutaneously (SC) once a week (QW) for 24 weeks.
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Placebo
Number analyzed (Participants) | 132 | 134 | 133
percentage of HbA1c | -1.34 (0.064) | -1.21 (0.064) | -0.54 (0.064)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-0.97 to -0.61]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-0.84 to -0.49]

2. Primary Outcome: Change From Baseline in the HbA1c at 24 Weeks (Efficacy Estimand)
Description: LS mean of the HbA1c change from baseline to primary endpoint at week 24 was adjusted by treatment, country, SGLT2 inhibitor dose, metformin use, treatment-by-visit interactions as fixed effects, and baseline HbA1c as a covariate and participant as a random effect, via a MMRM analysis. The efficacy estimand excluded post-rescue data and compared the benefit of randomized treatments when taken as directed without rescue medication.
Time Frame: Baseline, Week 24
Population: All randomized participants who received at least one dose of study drug and had a baseline and post-baseline value excluding values collected after rescue medication.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Placebo
Number analyzed (Participants) | 130 | 131 | 123
percentage of HbA1c | -1.33 (0.063) | -1.19 (0.063) | -0.51 (0.065)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.00 to -0.64]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-0.86 to -0.51]

3. Secondary Outcome: Percentage of Participants With HbA1c <7%
Description: Number of participants with an HbA1c value of <7% at Week 24 is measured using longitudinal logistic regression with repeated measurements. The model will include independent variables of treatment, country, SGLT2 inhibitor dose, metformin use, visit, treatment-by-visit interaction, and baseline HbA1c as a covariate.
Time Frame: 24 Weeks
Population: All participants who received at least one dose of Dulaglutide with HbA1c <7% at Week 24.
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Placebo
Number analyzed (Participants) | 142 | 141 | 140
percentage of participants
  Treatment-regimen Estimand: number analyzed (Participants) | 132 | 134 | 133
  Treatment-regimen Estimand | 71.21 | 60.45 | 31.58
  Efficacy Estimand: number analyzed (Participants) | 130 | 131 | 123
  Efficacy Estimand | 71.54 | 61.83 | 32.52
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Treatment-regimen Estimand; Test type: Superiority; p < .001, Regression, Logistic
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Placebo; Treatment-regimen Estimand; Test type: Superiority; p < .001, Regression, Logistic
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs Placebo; Efficacy Estimand; Test type: Superiority; p < .001, Regression, Logistic
Statistical Analysis 4: Comparison: 0.75 mg Dulaglutide vs Placebo; Efficacy Estimand; Test type: Superiority; p < .001, Regression, Logistic

4. Secondary Outcome: Change From Baseline in Body Weight at 24 Weeks
Description: LS mean of the body weight change from baseline to primary endpoint at week 24 was adjusted by treatment, country, SGLT2 inhibitor dose, metformin use, baseline HbA1c strata, treatment-by-visit interactions as fixed effects, and baseline body weight as a covariate and participant as a random effect, via a MMRM analysis
Time Frame: Baseline, Week 24
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Placebo
Number analyzed (Participants) | 142 | 141 | 140
kilograms (kg)
  Treatment-regimen Estimand: number analyzed (Participants) | 135 | 136 | 137
  Treatment-regimen Estimand | -3.1 (0.30) | -2.6 (0.30) | -2.1 (0.30)
  Efficacy Estimand: number analyzed (Participants) | 133 | 133 | 127
  Efficacy Estimand | -3.1 (0.30) | -2.6 (0.30) | -2.3 (0.31)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Treatment-regimen Estimand; Test type: Superiority; p = 0.027, Mixed Models Analysis; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.8 to -0.1]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Placebo; Treatment-regimen Estimand; Test type: Superiority; p = 0.264, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.3 to 0.4]
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs Placebo; Efficacy Estimand; Test type: Superiority; p = 0.059, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.7 to 0.0]
Statistical Analysis 4: Comparison: 0.75 mg Dulaglutide vs Placebo; Efficacy Estimand; Test type: Superiority; p = 0.435, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.2 to 0.5]

5. Secondary Outcome: Change From Baseline in Fasting Serum Glucose (Central Laboratory) at 24 Weeks
Description: LS mean of change from baseline was calculated using last observation carried forward (LOCF) by treatment group, adjusted for treatment, country, SGLT2 inhibitor dose, metformin use, baseline HbA1c strata, and baseline fasting serum glucose using analysis of covariance (ANCOVA).
Time Frame: Baseline, Week 24
Population: All participants who received at least one dose of study drug and had baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: milligram/deciliter (mg/dL)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Placebo
Number analyzed (Participants) | 142 | 141 | 140
milligram/deciliter (mg/dL)
  Treatment-regimen Estimand: number analyzed (Participants) | 134 | 133 | 132
  Treatment-regimen Estimand | -31.6 (2.17) | -26.5 (2.18) | -6.9 (2.21)
  Efficacy Estimand: number analyzed (Participants) | 132 | 130 | 122
  Efficacy Estimand | -31.9 (2.11) | -26.0 (2.12) | -5.3 (2.21)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Treatment-regimen Estimand; Test type: Superiority; p < .001, ANCOVA; Mean Difference (Final Values) = -24.7, 95% CI 2-sided [-30.8 to -18.6]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Placebo; Treatment-regimen Estimand; Test type: Superiority; p < 0.001, ANCOVA — Test was not controlled for type I error; Mean Difference (Final Values) = -19.6, 95% CI 2-sided [-25.7 to -13.5]
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs Placebo; Efficacy Estimand; Test type: Superiority; p < 0.001, ANCOVA — Test was not controlled for type I error; Mean Difference (Final Values) = -26.6, 95% CI 2-sided [-32.7 to -20.6]
Statistical Analysis 4: Comparison: 0.75 mg Dulaglutide vs Placebo; Efficacy Estimand; Test type: Superiority; p < 0.001, ANCOVA — Test was not controlled for type I error; Mean Difference (Final Values) = -20.7, 95% CI 2-sided [-26.7 to -14.6]

6. Secondary Outcome: Change From Baseline in 6-Point Self-Monitored Plasma Glucose (SMPG) Profile at 24 Weeks
Description: The self-monitored plasma glucose (SMPG) data were collected at the following 6 time points: pre-morning meal; 2 hours post-morning meal; pre-midday meal; 2 hours post-midday meal; pre-evening meal; 2 hours post-evening meal. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, metformin use, SGLT2 inhibitor use, country, visit, baseline HbA1c strata, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, Week 24
Population: All participants who received at least one dose of study drug and had baseline SMPG value and at least one post-baseline SMPG value.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Placebo
Number analyzed (Participants) | 142 | 141 | 140
mg/dL
  Pre-morning Morning Meal: number analyzed (Participants) | 128 | 124 | 128
  Pre-morning Morning Meal | -27.8 (2.13) | -23.2 (2.17) | -8.1 (2.14)
  2-Hour Postprandial Morning Meal: number analyzed (Participants) | 121 | 121 | 119
  2-Hour Postprandial Morning Meal | -44.6 (3.31) | -41.1 (3.30) | -20.1 (3.33)
  Pre-Mid Day Meal: number analyzed (Participants) | 127 | 124 | 126
  Pre-Mid Day Meal | -26.0 (2.91) | -22.0 (2.94) | -7.7 (2.93)
  2-Hour Postprandial Mid Day Meal: number analyzed (Participants) | 122 | 121 | 118
  2-Hour Postprandial Mid Day Meal | -31.8 (3.47) | -25.5 (3.47) | -12.8 (3.53)
  Pre-Evening Meal: number analyzed (Participants) | 128 | 121 | 124
  Pre-Evening Meal | -30.3 (2.85) | -30.1 (2.93) | -7.5 (2.91)
  2-Hour Postprandial Evening Meal: number analyzed (Participants) | 122 | 121 | 117
  2-Hour Postprandial Evening Meal | -36.0 (3.30) | -30.6 (3.31) | -13.9 (3.38)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Pre-morning meal; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -19.7, 95% CI 2-sided [-25.7 to -13.8]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Placebo; Pre-morning meal; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -15.2, 95% CI 2-sided [-21.2 to -9.2]
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs Placebo; 2-hour postprandial; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -24.5, 95% CI 2-sided [-33.8 to -15.3]
Statistical Analysis 4: Comparison: 0.75 mg Dulaglutide vs Placebo; 2-hour postprandial; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -21.1, 95% CI 2-sided [-30.3 to -11.8]
Statistical Analysis 5: Comparison: 1.5 mg Dulaglutide vs Placebo; Pre-midday meal; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -18.3, 95% CI 2-sided [-26.4 to -10.2]
Statistical Analysis 6: Comparison: 0.75 mg Dulaglutide vs Placebo; Pre-midday meal; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -14.3, 95% CI 2-sided [-22.5 to -6.2]
Statistical Analysis 7: Comparison: 1.5 mg Dulaglutide vs Placebo; 2-hour postprandial after midday meal; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -19.0, 95% CI 2-sided [-28.8 to -9.3]
Statistical Analysis 8: Comparison: 0.75 mg Dulaglutide vs Placebo; 2-hour postprandial after midday meal; Test type: Superiority; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = -12.8, 95% CI 2-sided [-22.5 to -3.1]
Statistical Analysis 9: Comparison: 1.5 mg Dulaglutide vs Placebo; Pre-evening meal; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -22.7, 95% CI 2-sided [-30.7 to -14.7]
Statistical Analysis 10: Comparison: 0.75 mg Dulaglutide vs Placebo; Pre-evening meal; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -22.5, 95% CI 2-sided [-30.7 to -14.4]
Statistical Analysis 11: Comparison: 1.5 mg Dulaglutide vs Placebo; 2-hour postprandial after evening meal; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -22.1, 95% CI 2-sided [-31.4 to -12.9]
Statistical Analysis 12: Comparison: 0.75 mg Dulaglutide vs Placebo; 2-hour postprandial after evening meal; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -16.7, 95% CI 2-sided [-26.0 to -7.4]

7. Secondary Outcome: Change From Baseline in Fasting Glucagon at 24 Weeks
Description: Change from baseline in fasting glucagon was analyzed using an ANCOVA model with last observation carried forward (LOCF) included in treatment, country, SGLT2i dose, metformin use, and baseline HbA1c strata as fixed effects and baseline fasting glucagon as a covariate (with and without post rescue data).
Time Frame: Baseline, Week 24
Population: All participants who received at least one dose of study drug and with non-missing baseline values and at least one post-baseline value at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: picomole per liter (pmol/L)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Placebo
Number analyzed (Participants) | 142 | 141 | 140
picomole per liter (pmol/L)
  Treatment-regimen Estimand | -2.1 (0.39) | -1.5 (0.39) | -0.9 (0.40)
  Efficacy Estimand: number analyzed (Participants) | 133 | 129 | 118
  Efficacy Estimand | -2.2 (0.39) | -1.4 (0.39) | -0.9 (0.41)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Treatment-regimen Estimand; Test type: Superiority; p = 0.032, ANCOVA; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.3 to -0.1]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Placebo; Treatment-regimen Estimand; Test type: Superiority; p = 0.273, ANCOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.7 to 0.5]
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs Placebo; Efficacy Estimand; Test type: Superiority; p = 0.023, ANCOVA; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-2.4 to -0.2]
Statistical Analysis 4: Comparison: 0.75 mg Dulaglutide vs Placebo; Efficacy Estimand; Test type: Superiority; p = 0.320, ANCOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.7 to 0.6]

8. Secondary Outcome: Rate of Hypoglycemic Events Adjusted Per 30 Days
Description: A hypoglycemic event is defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia, and has a PG level of ≤70 mg/dL (≤3.9 mmol/L).
Time Frame: Baseline through 24 Weeks
Population: All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Number of events/participant/30 days
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Placebo
Number analyzed (Participants) | 142 | 141 | 140
Number of events/participant/30 days
  Total Hypoglycemia | 0.026 (0.1827) | 0.022 (0.1375) | 0.017 (0.1320)
  Documented Symptomatic Hypoglycemia | 0.013 (0.1406) | 0.013 (0.1030) | 0.010 (0.0893)
  Asymptomatic Hypoglycemia | 0.013 (0.1180) | 0.008 (0.0639) | 0.006 (0.0540)
  Probable Symptomatic | 0.000 (0.0000) | 0.001 (0.0152) | 0.001 (0.0147)
  Relative Hypoglycemia | 0.003 (0.0311) | 0.001 (0.0150) | 0.005 (0.0493)
  Nocturnal Hypoglycemia | 0.002 (0.0288) | 0.009 (0.0821) | 0.000 (0.0000)

9. Secondary Outcome: Number of Participants Requiring Rescue Therapy Due to Severe Persistent Hyperglycemia
Description: Rescue therapy was defined as any additional therapeutic intervention in participants who developed persistent, severe hyperglycemia despite full compliance with the assigned therapeutic regimen, or initiation of an alternative antihyperglycemic medication following study drug discontinuation.
Time Frame: Baseline through 24 Weeks
Population: All participants who had at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Placebo
Number analyzed (Participants) | 142 | 141 | 140
Participants | 0 | 3 | 2

10. Secondary Outcome: Number of Participants With Adjudicated Acute Pancreatitis Events
Description: The number of participants with events of pancreatitis confirmed by adjudication were summarized cumulatively at 24 weeks. Pancreatitis events were adjudicated by a committee of physicians external to the Sponsor.
  A summary of serious and other non-serious events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 24 Weeks
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Placebo
Number analyzed (Participants) | 142 | 141 | 140
Participants | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Adjudicated Cardiovascular (CV) Events
Description: Death and selected nonfatal CV adverse events (AEs) were adjudicated by an independent committee of physicians with cardiology expertise external to the Sponsor. Nonfatal CV events that were to be adjudicated were myocardial infarction (MI); hospitalization for unstable angina; hospitalization for heart failure; coronary interventions such as coronary artery bypass graft (CABG) or ( percutaneous coronary intervention (PCI); and cerebrovascular events, including cerebrovascular accident (stroke) and transient ischemic attack (TIA).
Time Frame: Baseline through 24 Weeks
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Placebo
Number analyzed (Participants) | 142 | 141 | 140
Participants
  Any CV Event | 0 | 0 | 3
  Fatal CV Event | 0 | 0 | 0
  Non-fatal CV Event | 0 | 0 | 3

ADVERSE EVENTS:
Time Frame: Baseline to end of study (up to 24 weeks)
Description: All participants who received at least one dose of study drug.
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 2/142 | 0/141 | 0/140
Serious Adverse Events (participants affected / at risk) | 5/142 | 3/141 | 5/140
Other Adverse Events (participants affected / at risk) | 43/142 | 34/141 | 29/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1.5 mg Dulaglutide (N=142) | 0.75 mg Dulaglutide (N=141) | Placebo (N=140)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal cord injury lumbar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/65 (1) | 0/72 (0) | 0/74 (0)
Endometrial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/65 (1) | 0/72 (0) | 0/74 (0)
Malignant neoplasm of conjunctiva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/77 (1) | 0/69 (0) | 0/66 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mg Dulaglutide (N=142) | 0.75 mg Dulaglutide (N=141) | Placebo (N=140)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 14 (16) | 4 (5)
Nausea (Gastrointestinal disorders) | 21 (32) | 7 (13) | 5 (6)
Viral upper respiratory tract infection (Infections and infestations) | 9 (12) | 8 (10) | 11 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (15) | 12 (14) | 10 (14)
Headache (Nervous system disorders) | 8 (13) | 5 (8) | 13 (16)

LIMITATIONS AND CAVEATS:
One participant was randomized into the study but did not receive study drug. This participant was not included in the efficacy or safety analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol: GBGE (a) Protocol (2015-08-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT02597049/Prot_000.pdf
  • Study Protocol: GBGE (b) Protocol (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT02597049/Prot_001.pdf
  • Statistical Analysis Plan (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT02597049/SAP_002.pdf